CLINICAL TRIAL: NCT01192074
Title: Use of Ultrasound in Obstetric Neuraxial Analgesia and Anesthesia Data Base
Status: Terminated | Type: Observational
Why Stopped: Lack of personnel/research time to recruit participants.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 1147418
Record Dates: First submitted 2010-08-26; First posted 2010-08-31 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Pregnancy
Keywords: Obstetric; Analgesia; Anesthesia; Obstetric Anesthesia; Obstetric Analgesia; ultrasound; ultrasonography; epidural analgesia; epidural anesthesia; spinal anesthesia; neuraxial anesthesia; neuraxial analgesia; pregnancy; labor; cesarean delivery; cesarean section
MeSH Terms: conditions — Agnosia | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ultrasound of the spine: Pregnant women receiving labor epidural analgesia or spinal anesthesia for cesarean delivery
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Preprocedure ultrasound examination of the spine

SUMMARY:
This is a data base building project on the use of pre-procedure ultrasound for the performance of labor epidural pain relief and spinal anesthesia for cesarean deliveries. Data collection includes ultrasound measured depth, actual needle depth, angle of ultrasound probe, actual needle angle, success rates, patient height and weight, number of attempts needed to place the epidural needle or spinal needle. Currently we are looking at the agreement between ultrasound determined depth of the epidural space or intrathecal space with actual needle depth.

DETAILED DESCRIPTION:
All patients presenting in labor or are having a cesarean delivery are eligible except: patients who are under age 18, have contraindications to regional anesthesia, in advanced labor, having emergency conditions and/or unable to understand the consent process.

* Data collected include:
* Ultrasound depth in transverse and oblique sagittal views
* Actual needle depth
* Level of placement
* Number of separate needle placements
* Number of needle redirects
* Angle of probe
* Angle of needle
* Total number of attempts
* Pt height
* Pt weight
* Pt BMI
* Pt age
* Pt gravity/parity
* Pt co-morbidities, e.g. pre-eclampsia
* Procedure performed
* Operator (Attending, CA-1, CA-2, CA-3, CRNA)

What is currently being examined is the correlation between ultrasound depth of the target area vs actual needle depth

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in labor or scheduled for induction requesting labor epidural analgesia
* Pregnant women scheduled for cesarean delivery
* Pregnant women in labor who are going to have a non-emergent cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Emergency delivery
* Emergency cesarean section
* Advanced labor
* Contraindications to neuraxial analgesia/anesthesia
* Unable to understand consent
* Under the age of 18

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant patients in labor Pregnant patients scheduled for cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Correlation of Ultrasound vs Needle Depth | Beginning of ultrasound exam to end of ultrasound exam: average 5 min
  The ultrasound measured depth taken via oblique sagittal views and transverse views of the epidural space for epidural analgesia or intrathecal space for spinal anesthesia will be correlated with actual needle depth

SECONDARY OUTCOMES:
Attempt Number | Beginning of placement of epidural or spinal needle to end of placement: average 10 min
  The number of needle placement attemtps: an attempt is defined as a separate needle placement The number of needle redirects: a redirect is defined at the need for changing the angle of needle direction at each separate needle attempt

CONTACTS AND LOCATIONS:
Overall Officials: Steven T Fogel, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Women's and Children's Hospital, Columbia, Missouri, United States

REFERENCES:
- [Background] Carvalho JC. Ultrasound-facilitated epidurals and spinals in obstetrics. Anesthesiol Clin. 2008 Mar;26(1):145-58, vii-viii. doi: 10.1016/j.anclin.2007.11.007. PMID 18319185
- [Background] Arzola C, Davies S, Rofaeel A, Carvalho JC. Ultrasound using the transverse approach to the lumbar spine provides reliable landmarks for labor epidurals. Anesth Analg. 2007 May;104(5):1188-92, tables of contents. doi: 10.1213/01.ane.0000250912.66057.41. PMID 17456672
- [Background] Chin KJ, Perlas A, Singh M, Arzola C, Prasad A, Chan V, Brull R. An ultrasound-assisted approach facilitates spinal anesthesia for total joint arthroplasty. Can J Anaesth. 2009 Sep;56(9):643-50. doi: 10.1007/s12630-009-9132-8. Epub 2009 Jun 23. PMID 19548051
- [Background] Grau T, Bartusseck E, Conradi R, Martin E, Motsch J. Ultrasound imaging improves learning curves in obstetric epidural anesthesia: a preliminary study. Can J Anaesth. 2003 Dec;50(10):1047-50. doi: 10.1007/BF03018371. PMID 14656785
- [Background] Grau T, Leipold RW, Conradi R, Martin E. Ultrasound control for presumed difficult epidural puncture. Acta Anaesthesiol Scand. 2001 Jul;45(6):766-71. doi: 10.1034/j.1399-6576.2001.045006766.x. PMID 11421838